CLINICAL TRIAL: NCT01888744
Title: The Effect of the Type of Ovarian Stimulation Protocol on PGD Results: a Prospective Randomised Trial
Brief Title: Preimplantation Genetic Diagnosis (PGD) With Gonadotropin-releasing Hormone (GnRH) Agonist Versus Antagonist
Acronym: Avanti
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Christophe Blockeel, Professor Doctor, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/010
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Reproductive Endocrinology; Fertility; Optimal Stimulation Protocol
Keywords: Intracytoplasmic sperm injection (ICSI); PGD; GnrH agonist; GnRH antagonist
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; ganirelix; cetrorelix; Menotropins; Chorionic Gonadotropin; Progesterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (GnRH agonist group) (Active Comparator): The long GnRH agonist protocol starts on day 21 of the preceding cycle with the administration of GnRH agonist, Decapeptyl® 0,1 mg subcutaneously daily or buserelin acetate, Suprefact® 600 μg daily intranasal. The administration of highly purified human menopausal gonadotropin (hp-HMG), Menopur® 225 IU subcutaneously is started after three weeks of desensitization. The desensitization is checked by ultrasound (absence of cysts) and hormonal measurement (Estradiol levels < 80 pg/ml, FSH ≤ 10 IU/l and progesterone < 1,5ng/ml)
  Interventions: Drug: GnRH agonist; Drug: hP-hMG; Drug: Human chorionic gonadotropin; Drug: Progesterone
- Group 2 (GnRH antagonist group) (Active Comparator): Ovarian stimulation is started at day 2 of the menstrual cycle with 225 IU of HMG (Menopur ®) subcutaneously. At day 6 of the stimulation GnRH antagonist (Orgalutran®) 0,25 mg subcutaneously is added. Basal hormonal status will be confirmed in the antagonist group before starting.
  Interventions: Drug: GnRH antagonist; Drug: hP-hMG; Drug: Human chorionic gonadotropin; Drug: Progesterone

INTERVENTIONS:
Drug: GnRH agonist
  Other Names: Suprefact nasal spray
  Arms: Group 1 (GnRH agonist group)
Drug: GnRH antagonist
  Other Names: Orgalutran or Cetrotide
  Arms: Group 2 (GnRH antagonist group)
Drug: hP-hMG
  Other Names: Menopur
Drug: Human chorionic gonadotropin — induction of final oocyte maturation
  Other Names: Pregnyl
Drug: Progesterone
  Other Names: Utrogestan vaginal tablets

SUMMARY:
The aim of our study is to define the optimal ovarian stimulation protocol concerning PGD and for this reason we plan a randomized controlled trial (RCT) comparing gonadotropin-releasing hormone (GnRH) agonist protocol versus GnRH antagonist protocol. The follicle stimulating hormone (FSH) preparation in both arms will be highly purified FSH (Menopur®).

DETAILED DESCRIPTION:
Patients will be randomized at the outpatient clinic in two groups.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 39 years the day of oocyte retrieval
* BMI ≤ 29
* cycle rank 1
* menstrual cycle 25-36 days
* PGD or preimplantation genetic screening (PGS) requested
* ICSI
* Single embryo transfer (SET) on day 5

Exclusion Criteria:

* Polycystic Ovary Syndrome (PCOS) (according Rotterdam criteria)
* Hormonal disturbances
* Endometriosis grade III and IV

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of day 3 embryos for biopsy available | up to 6 weeks

SECONDARY OUTCOMES:
Number of mature cumulus-oocyte complexes | up to 6 weeks
clinical pregnancy rate | up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Reproductive Medicine, Brussels, Belgium